CLINICAL TRIAL: NCT01180595
Title: Randomized Control Study Using Roentgen Stereophotogrammetric Analysis (RSA) to Compare the Fixation of the Trabecular Metal Monoblock and the Trabecular Metal Modular Total Knee Arthroplasties
Brief Title: Roentgen Stereophotogrammetric Analysis (RSA) Trial Comparing Trabecular Metal Monoblock and Modular Tibial Components
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dalhousie University (Other)
Collaborators: Zimmer Biomet (Industry)
Responsible Party: Principal Investigator, Michael Dunbar, MD, PhD, Dalhousie University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDHA-RS/2011-010
Record Dates: First submitted 2010-08-11; First posted 2010-08-12 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; arthroplasty; knee joint; radiography; surgery; Bone Density; Outcome Assessment (Health Care)
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modular (Other): Trabecular Metal Modular Tibial Total Knee Component
  Interventions: Device: Trabecular Metal Modular Tibial Total Knee Component
- Monoblock (Other): Trabecular Metal Monoblock Tibial Total Knee Component
  Interventions: Device: Trabecular Metal Monoblock Tibial Total Knee Component

INTERVENTIONS:
Device: Trabecular Metal Modular Tibial Total Knee Component — The modular design of the Trabecular Metal Total Knee allows for increased options for physicians however, it is not clear how this modular feature will affect fixation since it may compromise some of the advantages of the original TM Monoblock tibial component.
  Arms: Modular
Device: Trabecular Metal Monoblock Tibial Total Knee Component
  Arms: Monoblock

SUMMARY:
Total knee replacement is an effective option for treating chronic knee conditions that cause pain and functional impairment. Significant improvements in quality of life, as measured by both disease specific and generic quality of life measures have been well documented. Carefully monitored introduction of new implant designs through small, randomized trials using radiostereometric analysis (RSA) is gaining support. RSA is a radiographic technique that uses small tantalum balls implanted into the patient's bone to measure micromotion (<1 mm) at the bone - implant interface, something which is not possible to do reliably using regular x-ray techniques. The amount of micromotion that occurs within 2 years of surgery can be used to predict the long term survival of knee replacements. This provides a method for detecting inferior implant designs using only a small number of patients before release of these products into large clinical trials.

The study purpose is to utilize RSA to compare the migration patterns of the Trabecular Metal(TM) Monoblock and the TM Modular Total Knee Arthroplasties during the first two postop years and to determine what proportion of cases achieve adequate fixation. Secondary outcome measures will be recorded to quantify changes in functional status of subjects after surgery and bone mineral density will be monitored to quantify any changes around the implant. Migration patterns will be compared to results obtained from previous studies of uncemented and cemented total knee arthroplasty components conducted at this centre.

Null Hypothesis: There is no significant difference in micromotion patterns of the TM arthroplasty components of the monoblock design and the modular design.

Alternative Hypothesis: There are significant differences in micromotion patterns between the tibial components of the monoblock design and the modular design.

This is a consecutive sample randomized control trial of patients undergoing total knee arthroplasty with the TM Monoblock and TM Modular Knee Arthroplasty systems utilizing RSA to identify the migration patterns of the tibial components of the implant. DEXA scanning will also be conducted to determine changes in the bone mineral density adjacent to the implant. Health status and functional outcome measures will be recorded to quantify functional status of subjects before surgery and at each follow-up interval. Gait will be monitored and analyzed preoperatively and postoperatively throughout the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic osteoarthritis of the knee indicating surgical intervention
* Between the ages of 21 and 80 inclusive
* Ability to give informed consent

Exclusion Criteria:

* Significant co-morbidity affecting ability to ambulate
* Flexion contracture greater than 15°
* Extension lag greater than 10°
* Tibial subluxation greater than 10 mm on standing AP radiograph
* Prior arthroplasty, patellectomy or osteotomy with the affected knee
* Lateral or medial collateral ligament instability (> 10° varus/valgus)
* Leg length discrepancy greater than 10 mm
* Active or prior infection
* Morbid Obesity (BMI > 40)
* Medical condition precluding major surgery
* Severe osteoporosis or osteopenia
* Neuromuscular impairment

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-02; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
micromotion of tibial component as measured with RSA | 2 years postoperative

SECONDARY OUTCOMES:
Bone mineral density around the tibial component | 2 years postoperative
Subjective health outcome questionnaires - SF36, WOMAC, Oxford12 knee, Pain and Catastrophizing Scale, Standardized comorbidity questionnaire | 2 years postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Dunbar, MD PhD, Principal Investigator — Dalhousie University and CDHA
Locations (1):
- Halifax Infirmary, Halifax, Nova Scotia, Canada